# Informed Consent Form (ICF)

# EFFECTIVENESS OF AN MHEALTH INTERVENTION, BASED ON REHABILITATION AND A PERSONALISED NUTRITION PLAN, IN THE RECOVERY AND IMPROVEMENT OF DYSPHAGIA IN PATIENTS DIAGNOSED WITH STROKE

Principal Investigator: Eduardo Sánchez-Sánchez

Principal Investigator Clinical Assistant Professor

Punta Europa University Hospital. Andalusian Healthcare

Service / Faculty of Nursing. University of Cadiz

Algeciras, Spain

Protocol identification number: AP-0331-2022-C3-F2

ClinicalTrials.gov identifier: NCT07267468 (started: 2025-11-13) (YYYY-MM-DD)

Authors of the ICF: Antonio-Jesús Marín-Paz & Eduardo Sánchez-Sánchez

Current state: - Approved by Cadiz Research Ethics Committee (143.22)

- Translation into English.

Version: 1.1 (2025-10-07)

### INFORMATION SHEET

Date: 2025-10-07

**Study Title:** Effectiveness of an mHealth intervention, based on rehabilitation and a personalised nutrition plan, in the recovery and improvement of dysphagia in patients diagnosed with stroke.

Principal Investigator: Eduardo Sánchez Sánchez

#### INTRODUCTION

You are invited to participate in a study which has been approved by the Clinical Research Ethics Committee of Cádiz.

Please read this information sheet carefully. The Investigator will clarify any doubts you may have.

# **VOLUNTARY PARTICIPATION**

Your participation in this study is voluntary and you may cancel your decision and withdraw your consent at any time without this altering your relationship with your nurse or your doctor, or causing prejudice to your treatment or the care you may require.

#### GENERAL DESCRIPTION OF THE STUDY

The study aims to evaluate the effectiveness of a mobile application (app) downloaded to your mobile phone for the improvement and recovery from difficulty swallowing liquids in patients who have suffered a stroke.

Should you have suffered a cerebrovascular accident and present with difficulty swallowing liquids, you may participate in this study.

You will be randomly selected for a group that receives general and routine care, or another group that will be provided with a mobile application (app) that you can download to your phone, where you will find information on nutritional, compensatory, and exercise measures related to this problem of swallowing liquids. As previously mentioned, assignment to one group or the other will be due to chance, without the investigators deciding which group you will belong to.

When you decide to participate in this research and are selected for a group, general, nutritional, and clinical data will be collected. Furthermore, you will be followed up at 3, 6, and 9 months, where data will continue to be collected to assess the effectiveness or otherwise of the mobile application and/or general measures.

The start of the study may take place in the hospital or upon discharge to your home/social and healthcare centre. This data will be collected through questionnaires, questions, ... and some body measurements. Clinical data will be collected through access to your Digital Clinical Record. This follow-up will be conducted by telephone, avoiding trips to the hospital centre.

# BENEFITS AND RISKS DERIVED FROM YOUR PARTICIPATION IN THE STUDY

The study aims to evaluate the effectiveness of a mobile application (app) downloaded to your mobile phone or any other device for the improvement and recovery from difficulty swallowing liquids in

patients who have suffered a stroke.

It is possible that this mobile application may not serve to improve or recover, beyond what is achieved through routine general and specific care.

Date: 2025-10-07

No adverse effects have been described with the use of mobile applications.

#### FINANCIAL COMPENSATION

Your participation in the study will not incur any cost to you, nor is there any financial compensation.

#### CONFIDENTIALITY

Your personal data collected during the performance of this study will be processed in accordance with the provisions of the European Union's General Data Protection Regulation (GDPR) and Organic Law 3/2018, of 5 December, on Personal Data Protection and Guarantee of Digital Rights (LOPDGDD).

The controller of personal data is: Eduardo Sánchez Sánchez. The contact details of the data controller are: phone: XXXXXXXXX and email: XXXXXXXX

The purpose of processing personal data is to conduct research.

Legal basis: the processing of personal data is covered by the legal basis established in Articles 6.1.a) and 9.2.a) of the GDPR, which establishes that processing will be lawful if the data subject or their legal representative has given explicit consent to the processing of their personal data for one or more specific purposes. The data subject or their legal representative may give their consent for the use of their personal data for health research purposes, and, in particular, biomedical research. The purpose may encompass categories related to general areas linked to a medical or research specialisation, all in accordance with the Seventeenth Additional Provision 2.a) of the LOPDGDD.

Recipients or categories of recipients. Your personal data will be treated with the utmost confidentiality and will therefore not be transferred to third parties outside the research project. There are no recipients or categories of recipients of your personal data. Your personal data will in no case be subject to an international transfer of personal data. If the results of the study are published, your personal data will not be published and your identity will remain anonymous.

# Exercise of personal data protection rights

You have the right to request from the controller access to your personal data undergoing processing. Likewise, you have the right to the rectification of your personal data, to the erasure of your personal data, to the restriction of processing, to object to processing, to data portability, and not to be subject to decisions based solely on the automated processing of your data, all in accordance with and within the limitations provided for in the GDPR and the LOPDGDD for health and biomedical research. These rights shall be exercised through the email address/postal address.

At any time, you may exercise the right to withdraw consent for the processing of your personal data, without affecting the lawfulness of processing for health research purposes based on consent given prior to its withdrawal. This right shall be exercised through the email address/postal address.

You have the right to lodge a complaint with the supervisory authority, which is the Council for Transparency and Personal Data Protection of Andalusia, which exercises its competence over the processing of personal data managed by the autonomous institutions of Andalusia, by the autonomous administration, by local administrations, and by other public and private law entities dependent on any of them, as well as by the universities of the Andalusian university system. For all other cases, you have the right to lodge a complaint with the Spanish Data Protection Agency.

Date: 2025-10-07

#### **FUNDING**

**Signatures:** 

This study has competitive public funding through the FPS2020 call for R&D&I Projects in Primary Care, Regional, and CHARES centres.

#### WITHDRAWAL OF CONSENT

You may withdraw your consent at any time without having to give explanations. You should also know that you may be excluded from the study if the study investigators deem it appropriate. You have the right to be informed of any changes to the study. In that case, the investigator will have to ask you for new consent, which you would be entitled to refuse.

Before signing, please read the document carefully, ask all the questions you consider appropriate, and if you wish, consult it with all the people you deem necessary. In case of doubt, you should contact the Principal Investigators, David Sánchez Relinque and María Eugenia Valenzuela Mateos.

| Participant's Signature: |
|---------------------------|
| Name: |
| Date: |
| Investigator's Signature: |
| Name: |
| Data |

# WRITTEN INFORMED CONSENT

Date: 2025-10-07

**Study Title:** Effectiveness of an mHealth intervention, based on rehabilitation and a personalised nutrition plan, in the recovery and improvement of dysphagia in patients diagnosed with stroke.

| Sponsor: Eduardo Sánchez Sánchez | |
|---|---|
| (full name) | |
| <ul> <li>I have read and understood the information sheet provided to me.</li> <li>I have been able to ask questions about the study.</li> </ul> | |
| • I have received sufficient information about the study. I have spoken with: | |
| (name of the investigator | r) |
| understand that my participation is voluntary. I understand that I can withdraw from the st | udy: |
| • At any time. | |
| • Without having to give explanations. | |
| <ul> <li>Without this affecting my medical care.</li> </ul> | |
| freely give my consent to participate in the study. | |
| DATE: | |

PARTICIPANT'S SIGNATURE

# ORAL CONSENT BEFORE WITNESSES

**Study Title:** Effectiveness of an mHealth intervention, based on rehabilitation and a personalised nutrition plan, in the recovery and improvement of dysphagia in patients diagnosed with stroke.

Date: 2025-10-07

| Sponsor: Eduardo Sánchez Sánchez | |
|---|---|
| Iresponsibility that | (full name), declare on my own (name of the study participant) |
| <ul> <li>Has received the study information sheet.</li> <li>Has been able to ask questions about the study.</li> <li>Has received sufficient information about the study.</li> <li>Has been informed by:</li> </ul> | |
| (name of the investigator) | |

Understands that their participation is voluntary. They understand that they can withdraw from the study:

- At any time.
- Without having to give explanations.
- Without this affecting their medical care.

And has freely expressed their consent to participate in the study.

WITNESS'S SIGNATURE

# REPRESENTATIVE'S CONSENT

Date: 2025-10-07

**Study Title:** Effectiveness of an mHealth intervention, based on rehabilitation and a personalised nutrition plan, in the recovery and improvement of dysphagia in patients diagnosed with stroke.

| | | (full name) |
|---|---|---|
| in my | | (relationship to the participant) of (name of the study participant) |
| • | I have read and understood the st<br>I have been able to ask questions<br>I have received satisfactory answ<br>I have received sufficient informations<br>I have spoken with: | about the study. ers to my questions. |
| | | (name of the investigator) |
| I unde | rstand that participation is voluntar | y. I understand that they can withdraw from the study: |
| • | At any time. Without having to give explanation Without this affecting their media | |
| In my<br>been g | presence,iven all relevant information adapt | (name of the study participant) has ed to their level of understanding and agrees to participate. |
| | give my consent foricipate in this study. | (name of the study participant) |
| DATE | /• | |

REPRESENTATIVE'S SIGNATURE

# HOJA DE INFORMACIÓN

Fecha: 2025-10-07

**Título del estudio:** Efectividad de una intervención de mHealth, basado en la rehabilitación y plan de nutrición personalizado, en la recuperación y mejora de la disfagia en pacientes con diagnóstico de accidente cerebrovascular.

Investigador principal: Eduardo Sánchez Sánchez

## INTRODUCCION

| Se le invita a particip | ar en un | estudio | que ha | sido | aprobado por | el Comité | Ético de Inv | estigación |
|---|---|---|---|---|---|---|---|---|
| Clínica de Cádiz. Por | favor, | lea | esta | hoja | informativa | a con | atención. | |
| El investigador | | | | | le aclarará | i las dudas | que le puedar | ı surgir. |

#### PARTICIPACIÓN VOLUNTARIA

Su participación en este estudio es voluntaria y usted puede anular su decisión y retirar el consentimiento en cualquier momento sin que por ello se altere su relación con la enfermera o con su doctora ni se produzca perjuicio en su tratamiento o en la atención que usted pueda necesitar.

#### DESCRIPCIÓN GENERAL DEL ESTUDIO

El estudio pretende evaluar la eficacia de una aplicación móvil que se descarga en su teléfono móvil para la mejora y recuperación de la dificultad para tragar líquidos en pacientes que han sufrido un accidente cerebrovascular.

En caso de que usted haya sufrido un accidente cerebrovascular y presenta dificultad para tragar líquidos, podrá participar en este estudio. Mediante el azar será seleccionado para un grupo que recibe los cuidados generales y habituales u otro grupo al que se le proporcionará una aplicación móvil para que se la pueda descargar en su móvil y donde podrá tener información sobre medidas nutricionales, compensatorias y de ejercicio relacionadas con este problema al tragar líquidos. Tal y como hemos mencionado con anterioridad, la pertenencia a un grupo u otro será debido al azar, sin que los investigadores decidan a qué grupo pertenecerá.

Cuando usted decida participar en esta investigación y se seleccione para un grupo se recogerán datos generales, nutricionales, clínicos, ... Además, se le realizará un seguimiento a los 3, 6 y 9 meses, donde se seguirán recogiendo datos para valorar la eficacia o no de la aplicación móvil y/o medidas generales. El inicio del estudio se puede realizar en el hospital o al alta a su domicilio/centro sociosanitario.

Estos datos se recogerán mediante cuestionarios, preguntas, ... y algunas medidas corporales. Los datos clínicos serán recogidos gracias al acceso a su Historia Clínica Digital. Este seguimiento será telefónico, evitando traslados al centro hospitalario.

### BENEFICIOS Y RIESGOS DERIVADOS DE SU PARTICIPACIÓN EN EL ESTUDIO

El estudio pretende evaluar la eficacia de una aplicación móvil que se descarga en su teléfono móvil o cualquier otro dispositivo para la mejora y recuperación de la dificultad para tragar líquidos en pacientes que han sufrido un accidente cerebrovascular. Es posible que esta aplicación móvil no sirva para mejorar o recuperarse, más allá del obtenido a través de los cuidados generales y específicos rutinarios.

No se han descrito efectos adversos en el uso de aplicaciones móviles.

# COMPENSACIÓN ECONÓMICA

Su participación en el estudio no supondrá ningún gasto para usted, ni existe compensación económica.

Fecha: 2025-10-07

#### CONFIDENCIALIDAD

Sus datos personales recogidos en la realización de este estudio serán tratados según lo establecido en el Reglamento General de Protección de Datos de la Unión Europea (RGPD) y la Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos de Carácter Personal y garantía de los derechos digitales (LOPDGDD).

El responsable del tratamiento de datos personales es: Eduardo Sánchez Sánchez. Los datos de contacto del responsable de tratamiento son: tfno.: XXXXXXXX y correo electrónico: XXXXXXXXXX

La finalidad del tratamiento de datos personales es la realización de una investigación.

Base legal: el tratamiento de datos personales se encuentra amparado en la base legal establecida en los arts. 6.1.a) y 9.2.a) del RGPD, que establece que el tratamiento será lícito si el interesado o su representante legal dio su consentimiento explícito para el tratamiento de sus datos personales para uno o varios fines específicos.

El interesado o su representante legal puede otorgar su consentimiento para el uso de sus datos personales con fines de investigación en salud, y, en particular, la biomédica.

La finalidad puede abarcar categorías relacionadas con áreas generales vinculadas a una especialidad médica o investigadora, todo ello de conformidad con la Disposición adicional decimoséptima 2.a) de la LOPDGDD.

Destinatarios o categorías de destinatarios. Sus datos personales serán tratados con la más absoluta confidencialidad por lo que no serán cedidos a terceras personas ajenas al proyecto de investigación. No existen destinatarios o categorías de destinatarios de sus datos personales. En ningún caso sus datos personales van a ser objeto de una transferencia internacional de datos personales. Si se publican los resultados del estudio, sus datos personales no serán publicados y su identidad permanecerá anónima.

# Ejercicio de los derechos de protección de datos personales.

Tiene derecho a solicitar al responsable el acceso a sus datos personales sometidos a tratamiento. Asimismo, tiene derecho a la rectificación de sus datos personales, a la supresión de sus datos personales, a la limitación del tratamiento, a oponerse al tratamiento, a la portabilidad de los datos y a no ser objeto de decisiones basadas únicamente en el tratamiento automatizado de sus datos, todo ello de conformidad y con las limitaciones previstas en el RGPD y en la LOPDGDD para la investigación en salud y biomédica. Estos derechos se ejercerán a través de la dirección de correo electrónico/dirección postal.

En cualquier momento puede ejercer el derecho a retirar el consentimiento para el tratamiento de sus datos personales, sin que ello afecte a la licitud del tratamiento con fines de investigación sanitaria basado en el consentimiento previo a su retirada. Este derecho se ejercerá a través de la dirección de correo electrónico/dirección postal.

Tiene el derecho a presentar una reclamación ante la autoridad de control, que es el Consejo de Transparencia y Protección de Datos Personales de Andalucía, que ejercer su competencia para los tratamientos de datos personales gestionados por las instituciones autonómicas de Andalucía, por la Administración autonómica, por las Administraciones locales, y por otras entidades de derecho

público y privado dependientes de cualquiera de ellas, así como por las universidades del sistema universitario andaluz. Para el resto de los supuestos tiene el derecho a presentar una reclamación ante la Agencia Española de Protección de Datos.

Fecha: 2025-10-07

# FINANCIACIÓN

Este estudio dispone de financiación pública competitiva a través de la convocatoria FPS2020-Proyectos de I+i en atención primaria, comarcales y CHARES.

# RETIRADA DEL CONSENTIMIENTO

Usted puede retirar su consentimiento en cualquier momento sin tener que dar explicaciones.

También debe saber que puede ser excluido del estudio si los investigadores del estudio lo consideran oportuno.

Usted tiene derecho a estar informado de cualquier cambio en el estudio. En ese caso, el investigador tendrá que pedirle un nuevo consentimiento que usted podría rechazar.

Antes de firmar, lea detenidamente el documento, haga todas las preguntas que considere oportunas, y si lo desea, consúltelo con todas las personas que considere necesario. En caso de duda debe dirigirse a los investigadores principales, David Sánchez Relinque y María Eugenia Valenzuela Mateos

| Firmas:<br>Firma del paciente: | Firma del Investigador: |
|--------------------------------|-------------------------|
| Nombre: | Nombre: |
| Fecha: | Fecha: |

de accidente cerebrovascular.

FECHA:

Promotor: Eduardo Sánchez Sánchez

Fecha: 2025-10-07

**Título del estudio:** Efectividad de una intervención de mHealth, basado en la rehabilitación y plan de nutrición personalizado, en la recuperación y mejora de la disfagia en pacientes con diagnóstico

| Yo (nomb | ore y apellidos) |
|---|---|
| | He leído y comprendido la hoja de información que se me ha entregado. He |
| | podido hacer preguntas sobre el estudio. |
| | He recibido suficiente información sobre el estudio. He |
| | hablado con: |
| | (nombre del investigador) |
| | Comprendo que mi participación es voluntaria. Comprendo |
| | que puedo retirarme del estudio: |
| | 1º Cuando quiera |
| | 2° Sin tener que dar explicaciones. |
| | 3º Sin que esto repercuta en mis cuidados médicos. |
| | Presto libremente mi conformidad para participar en el estudio. |

FIRMA DEL PARTICIPANTE

FECHA:

# **CONSENTIMIENTO ORAL ANTE TESTIGOS**

**Título del estudio:** Efectividad de una intervención de mHealth, basado en la rehabilitación y plan de nutrición personalizado, en la recuperación y mejora de la disfagia en pacientes con diagnóstico de accidente cerebrovascular.

| o (nombre y apellidos) | declaro bajo mi responsabilidad qu |
|---|---|
| | (nombre del participante en el estudio) |
| Ha recibido la hoja de informa | ación sobre el estudio. |
| Ha podido hacer preguntas sol | bre el estudio. |
| Ha recibido suficiente informa | ación sobre el estudio. |
| Ha sido informado por: | |
| Comprende que su participacione que puede retirarse del estudio | • |
| que puede retirarse del estudio | • |
| 10 Cuanda aviana | |
| 1º Cuando quiera. | |
| 2° Sin tener que dar explicacion | ones. |
| • | |

FIRMA DEL TESTIGO

# CONSENTIMIENTO DEL REPRESENTANTE

**Título del estudio:** Efectividad de una intervención de mHealth, basado en la rehabilitación y plan de nutrición personalizado, en la recuperación y mejora de la disfagia en pacientes con diagnóstico de accidente cerebrovascular.

| Promotor: Eduardo Sánchez Sánchez |
|---|
| Yo (nombre y apellidos)en calidad de |
| (relación con el participante) de(nombre del participante en |
| estudio) |
| He leído y comprendido la hoja de información sobre el estudio.<br>He podido hacer preguntas sobre el estudio. |
| He recibido respuestas satisfactorias a mis preguntas. |
| He recibido suficiente información sobre el estudio. |
| He hablado con: |
| (nombre del investigador) |
| Comprendo que la participación es voluntaria. |
| Comprende que puede retirarse del estudio: |
| 1º Cuando quiera. |
| 2° Sin tener que dar explicaciones. |
| 3° Sin que esto repercuta en sus cuidados médicos. |
| En mi presencia se ha dado a(nombre del participante en el |
| estudio) toda la información pertinente adaptada a su nivel de entendimiento y está de |
| acuerdo en participar. |
| Y presto mi conformidad con que(nombre del participante en |
| el estudio) participe en este estudio. |
| FECHA: FIRMA DEL REPRESENTANTE |